CLINICAL TRIAL: NCT03535558
Title: Fluoroquinolone Associated Disability
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108484; RRA-20379 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Bronchitis; Sinusitis; Urinary Tract Infections
MeSH Terms: conditions — Bronchitis; Sinusitis; Urinary Tract Infections | interventions — Fluoroquinolones; Azithromycin; Sulfamethoxazole; Trimethoprim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: FQ With Uncomplicated Sinusitis or Bronchitis: A target cohort which includes participants exposed to an oral fluoroquinolone (FQ) with an occurrence start between 2007-01-01 and 2015-12-31 (inclusive) and are between 18 and 65 years of age (inclusive). All participants must have continuous observation of at least 180 days prior and 120 days after event index date, and all events will be evaluated per participant. The members of the treatment groups will be linked to the Truven Health and Productivity Management (HPM) data set.
  Interventions: Drug: Fluoroquinolone (FQ)
- Cohort 2: FQ With Uncomplicated Acute Urinary Tract Infection: A target cohort which includes participants exposed to an oral sulfamethoxazole/trimethoprim (ST) with a qualifying indication of uncomplicated acute urinary tract infection and an occurrence start between 2007-01-01 and 2015-12-31 (inclusive) and are between 18 and 65 years of age (inclusive). All participants must have continuous observation of at least 180 days prior and 120 days after event index date, and all events will be evaluated per participant. The members of the comparator groups will be linked to the Truven HPM data set.
  Interventions: Drug: Fluoroquinolone (FQ)
- Cohort 3: AZ with Uncomplicated Acute Sinusitis or Bronchitis: A comparator cohort which includes participants exposed to oral azithromycin (AZ) with a qualifying indication of uncomplicated acute sinusitis or bronchitis and an occurrence start between 2007-01-01 and 2015-12-31 (inclusive) and are between 18 and 65 years of age (inclusive). All participants must have continuous observation of at least 180 days prior and 120 days after event index date, and all events will be evaluated per participant. The members of the comparator groups will be linked to the Truven HPM data set.
  Interventions: Drug: Azithromycin (AZ)
- Cohort 4: ST with Uncomplicated Acute Urinary Tract Infection: A comparator cohort which includes participants exposed to oral sulfamethoxazole/trimethoprim (ST) with a qualifying indication of uncomplicated acute urinary tract infection and an occurrence start between 2007-01-01 and 2015-12-31 (inclusive) and are between 18 and 65 years of age (inclusive). All participants must have continuous observation of at least 180 days prior and 120 days after event index date, and all events will be evaluated per participant. The members of the treatment groups will be linked to the Truven Health and Productivity Management (HPM) data set.
  Interventions: Drug: Sulfamethoxazole/Trimethoprim (ST) Fixed Dose Combination

INTERVENTIONS:
Drug: Fluoroquinolone (FQ) — Participants exposed to an oral FQ will be observed. The oral FQ included are Levofloxacin, Ciprofloxacin, Moxifloxacin, Ofloxacin, Gemifloxacin. Participants will not receive any intervention as a part of this study.
  Groups: Cohort 1: FQ With Uncomplicated Sinusitis or Bronchitis; Cohort 2: FQ With Uncomplicated Acute Urinary Tract Infection
Drug: Azithromycin (AZ) — Participants exposed to an oral AZ will be observed. Participants will not receive any intervention as a part of this study.
  Groups: Cohort 3: AZ with Uncomplicated Acute Sinusitis or Bronchitis
Drug: Sulfamethoxazole/Trimethoprim (ST) Fixed Dose Combination — Participants exposed to an oral ST will be observed. Participants will not receive any intervention as a part of this study.
  Groups: Cohort 4: ST with Uncomplicated Acute Urinary Tract Infection

SUMMARY:
The purpose of this study is to: 1) describe drug utilization for Fluoroquinolone(FQ), Azithromycin (AZ) and Sulfamethoxazole/Trimethoprim(ST) in the entire Truven MarketScan Commercial Claims and Encounters database (CCAE) database, and specifically among individuals in the Health and Productivity Management (HPM) during the observation period; 2) describe the rate of disability associated with 2 or more System Organ Class adverse events (SOC AEs) and exposure to FQs for several acute, uncomplicated indications; and 3) compare the rates of disability for 2 or more SOC AEs and exposure to FQs and AZ/ST for the same indications.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the Truven CCAE database who were eligible for disability insurance and can be linked to the Truven Health and Productivity Management (HPM) database
* Study participants will be included if they have 6 months of history before the first day on FQ or AZ/ST and at least 120 days afterward

Exclusion Criteria:

* If any protocol specified medical conditions or exposure to the protocol specified medications in the 6 months preceding the first qualifying dose of FQ or AZ/ST
* If participants have any disability claim in the 6 months preceding the qualifying FQ or AZ/ST dose
* If participants have the protocol specified condition-specific diagnoses within the 3 months preceding the qualifying FQ or AZ/ST exposure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants in the Truven Commercial Claims and Encounters (CCAE) database who were eligible for disability insurance and can be linked to the Truven HPM database. The study population will include individuals who had uncomplicated acute bacterial sinusitis, or bronchitis and were prescribed an oral fluoroquinolone (FQ) or oral azithromycin(AZ) and sulfamethoxazole/trimethoprim (ST) for urinary tract infection.
Sampling Method: Probability Sample
Enrollment: 239306 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Disability in Temporal Proximity | Up to 120 days
  Number of participants with disability in temporal proximity to 2 confirmed System Organ Class (SOC) adverse event (AEs) among the 6 of interest (peripheral nervous system, neuropsychiatric, musculoskeletal, sensory, cardiovascular, skin) will be reported. Disability is defined as an incident short-term disability claim in the Health and Productivity Management (HPM) database if it is observed within 120 days of the first Fluoroquinolone(FQ) or Azithromycin/ Sulfamethoxazole/Trimethoprim (AZ/ST) exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development,LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Janssen Investigative Site, Titusville, New Jersey, United States